CLINICAL TRIAL: NCT05523856
Title: Comparative Effectiveness of New Treatment Modalities for Localized Prostate Cancer
Brief Title: New Treatment Modalities for Localized Prostate Cancer
Acronym: TTOPROST/OBS
Status: Active, not recruiting | Type: Observational
Sponsor: Fundacion IMIM (Other)
Collaborators: Hospital Universitari de Bellvitge (Other); Institut d'Investigació Biomèdica de Bellvitge (Other); Hospitales Universitarios Virgen del Rocío (Other); Hospital Regional Universitario Carlos Haya (Other); Hospital del Mar (Other); Hospital Universitario Rey Juan Carlos (Other); Hospital Provincial de Castellon (Other); Hospital Arnau de Vilanova (Other); Hospital Universitario La Paz (Other); Hospital Universitario La Fe (Other); Hospital de Meixoeiro (Other Government); Hospital Universitario 12 de Octubre (Other); Hospital Universitario Reina Sofia de Cordoba (Other Government); Hospital General Universitario de Valencia (Other)
Responsible Party: Principal Investigator, Montserrat Ferrer, Medical Doctor, PhD, Fundacion IMIM
Other Study IDs: PI15/00296
Record Dates: First submitted 2022-07-26; First posted 2022-08-31 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
Keywords: Prostatic neoplasms; Active Surveillance; Robot-assisted radical prostatectomy; Intensity-Modulated Radiotherapy; Real-time brachytherapy; Health-related quality of life; Patient-Reported Outcomes; PRO; Impact; Comparative effectiveness research
MeSH Terms: conditions — Prostatic Neoplasms; Tooth, Impacted | interventions — Watchful Waiting; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- New Treatment Modalities Cohort: A consecutive sample of clinically localized prostate cancer patients treated with active surveillance, robot-assisted radical prostatectomy, intensity-modulated radiotherapy, or real-time brachytherapy in 18 Spanish hospitals.
  Interventions: Procedure: Active Surveillance; Procedure: Robot-Assisted Radical Prostatectomy; Radiation: Intensity-Modulated Radiotherapy; Radiation: Real-time brachytherapy

INTERVENTIONS:
Procedure: Active Surveillance — It consists on monitoring the cancer with regular tests including PSA, blood test and digital rectal examination every 6 months, a magnetic resonance imaging and prostate biopsy at the first year, and based on clinical decision thereafter. If there was a change on the results, the patient is considered for treatment.
Procedure: Robot-Assisted Radical Prostatectomy — It consists on the removal of the prostate gland and seminal vesicles with neurovascular preservation whenever anatomically and oncologically possible, with the Da Vinci procedure. Access is made through 5 or 6 small incisions, less than 1 cm. An extended pelvic lymph node dissection is performed when the risk estimation of node involvement is above the 5%. After surgery, the patient will be hospitalized for about 3 days and will probably resume his work activity between 3 and 5 weeks.
Radiation: Intensity-Modulated Radiotherapy — Patients in this group undergo volumetric modulated arc therapy under daily image-guided radiation therapy in the supine position. Radiation is delivered in 2-3 Gy daily fractions, 5 days per week, with a prescription dose of 60-70 Gy to the prostate.
Radiation: Real-time brachytherapy — Patients in this group receive I125 permanent seeds (low dose rate). The images are obtained with a transrectal ultrasound probe and are transferred to a planning system for calculating the number and position of the seeds. The prescrption dose is 145 Gy to the reference isodose (100%).

SUMMARY:
The purpose of this study is to evaluate the effectiveness of four of the nowadays most established primary treatments for patients with clinically localized prostate cancer (active surveillance, robot-assisted radical prostatectomy, intensity-modulated radiotherapy, and real-time brachytherapy) at short-, mid- and long-term follow-up. The primary aim is assessing the impact of treatments' side effects on patient's quality of life. As secondary objectives, biochemical disease-free survival, overall survival, and prostate cancer-specific survival will also be assessed.

DETAILED DESCRIPTION:
Primary Objective:

To compare the impact of active surveillance, robot-assisted radical prostatectomy, intensity-modulated radiotherapy, and real-time brachytherapy in patients with localized prostate cancer, in Patient-Reported Outcome Measures, considering side effects and physical and mental health at short-, mid- and long-term follow-up.

Secondary Objectives:

To assess biochemical disease-free survival by treatment and risk group, at mid- and long-term follow-up.

To assess overall survival by treatment and risk group, at mid- and long-term follow-up.

To assess prostate cancer-specific survival by treatment and risk group, at mid- and long-term follow-up.

To assess perceived general health and cancer-specific quality of life by treatment and risk group, at short-, mid- and long-term follow-up.

To assess benefits and risks of the new treatment modalities for localized prostate cancer, compared with the traditional ones (open radical prostatectomy, external-beam radiotherapy and intersticial pre-planned brachytherapy).

To assess utilities with direct and indirect methods.

Outline:

This is a prospective observational study of a cohort with clinically localized prostate cancer treated with either active surveillance, robot-assisted radical prostatectomy, intensity-modulated radiotherapy, or real-time brachytherapy.

Participants are consecutively recruited in 18 Spanish hospital departments (located in six autonomous communities). Patients eligible for inclusion were: age 50-75, tumor stage T1c or T2a, N0 and M0; Gleason ≤ 6 (or 3+4 if T1c); Prostate Specific Antigen (PSA) ≤ 10 ng/mL; and to be treated with active surveillance, robot-assisted radical prostatectomy, intensity-modulated radiotherapy, or real-time brachytherapy. Patients were excluded when body mass index was >33, they had undergone neoadjuvant hormonal treatment, previous pelvic treatments, and/or had presence of serious comorbidities. The decision regarding treatment is made jointly by patients and health professionals.

Demographic and clinical characteristics at baseline are recorded at clinical sites and include age, PSA, Gleason score, prostate volume, risk group and use of adjuvant hormonal treatment. According to the national health guidelines, participants will be visited every 6-12 months after treatment, and at least annualy thereafter.

Quality of Life questionnaires are administered centrally by telephone interview before treatment and during follow-up at 1, 3, 6, and 12 months after treatment the first year, and annually thereafter. Quality of Life evaluations are gathered using computer-assisted telephone administration and include: (1) the Expanded Prostate cancer Index Composite (EPIC), specifically designed to measure the impact of the different treatments; (2) 36-item Short-Form Health Survey version 2 (SF-36v2); (3) the EuroQol-5 Dimension (EQ-5D-5L); and (4) the Patient-Oriented Prostate Utility Scale (PORPUS).

The sample size calculated to detect small differences between groups (0.3 SD) on the EPIC or SF-36v2 scores was of 90 patients per treatment group, given a statistical power of at least 80% at a significance level of 5%, and loss to follow-up of 10%.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 75 years.
* Clinical stage T1 or T2, N0/Nx and M0/Mx.
* Gleason ≤6 or 7 (if 3+4 with T1c).
* Prostate-Specific Antigen (PSA) ≤ 10 .
* To be treated with active surveillance, robot-assisted radical prostatectomy, intensity-modulated radiotherapy or real-time brachytherapy

Exclusion Criteria:

* Body mass index > 33.
* Neoadjuvant hormonal treatment.
* Previous pelvic treatments.
* Presence of serious comorbidities.

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinically localized prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Impact of treatments' side effects on patients' quality of life measured in terms of change in the score of the Expanded Prostate Cancer Index Composite (EPIC) from baseline to 1, 3, 6, 12, 24, 60, 84, 120, 180, and 240 months after treatment. | Baseline to 1, 3, 6, 12, 24, 60, 84, 120, 180, and 240 months after treatment
  The Expanded Prostate Cancer Index Composite-26 (EPIC-26) is a prostate cancer-specific questionnaire that measures urinary, sexual, bowel, and hormonal domains, ranging from 0 to 100. Response options for each EPIC item are on a 4-, 5-, or 6-level Likert scale. Items are grouped in summary scores for sexual, bowel, and hormonal domains, and in 2 scores for the urinary domain (incontinence and irritative/obstructive symptoms), which are transformed linearly to a scale from 0 to 100, where higher scores indicate better outcomes.

SECONDARY OUTCOMES:
Biochemical disease-free survival | 5, 7, 10, 15, and 20 years after treatment
  Number of participants who are free of biochemical relapse after a specified duration of time. Biochemical relapse is measured by PSA levels. For patients treated with radical prostatectomy, biochemical relapse criteria of the American Urological Association is applied, and for patients treated with external radiotherapy or brachytherapy, criteria of the American Society for Therapeutic Radiology and Oncology is followed.
Overall survival | 5, 7, 10, 15, and 20 years after treatment
  Number of participants who are alive after a specified duration of time. Vital status and data of death from any cause recorded by linkage with the National Institute of Statistics.
Prostate cancer-specific survival | 5, 7, 10, 15, and 20 years after treatment
  Number of participants who are not dead due to prostate cancer after a specified duration of time. Death due to prostate cancer according to the cause of death registered in the the National Institute of Statistics.
Perceived general health measured with the 36-item Short-Form Health Survey version 2 (SF-36v2) | Baseline to 1, 3, 6, 12, 24, 60, 84, 120, 180, and 240 months after treatment
  The 36-Item Short-Form Health Survey version 2 (SF-36v2) contains 36 items covering eight dimensions: physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems and mental health. For each dimension, a score ranges from 0-100 (higher score indicate better health).Physical and mental component summaries are constructed, using recommended scoring algorithms. Summary scores are standardized to have a mean of 50 and standard deviation of 10 in the US general population.
Quality-Adjusted Life Years measured with the EuroQol-5 Dimensions | Baseline to 1, 3, 6, 12, 24, 60, 84, 120, 180, and 240 months after treatment
  The EuroQol-5 Dimensions (EQ-5D-5L) is a generic econometric instrument that contains five dimensions of health (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) with five levels of severity in each dimension. From the possible combinations of scales and severity levels (3125 health states), a utility index is obtained, which ranges from 1 (perfect health) to negative values, 0 being the value attributed to death.
Disease-specific Quality-Adjusted Life Years measured with the Patient-Oriented Prostate Utility Scale | Baseline to 1, 3, 6, 12, 24, 60, 84, 120, 180, and 240 months after treatment
  The Patient-Oriented Prostate Utility Scale (POPRUS) is a 10-attribute health state classification system that includes 5 broad items of health-related quality of life (pain, energy, social support, communication with doctor, and emotional well-being) and 5 prostate cancer-specific items (urinary frequency and incontinence, sexual function and desire, and bowel function. A multiattribute utility function is constructed using the patient-weighted utilities elicited with standard gamble. This utility index (PORPUS-U) ranges from 1 (perfect health) to 0 (dead).

IPD SHARING:
Plan to Share IPD: Yes
Data processing complies with ethical principles and relevant national and international legislation (Reglamento General de Protección de Datos 2016/679 and Organic Law 3/2018, of December 5). The final data will only be accessible to people working on the study. No data used in the analyses and subsequent dissemination of the study results will contain any identifiable reference referring to the names of patients. Once the study is finished, the results will be communicated to the competent authorities, in accordance with local legislation.
  Data and associated documentation will be made available to users only under a data sharing agreement that provides for:
  * A commitment to use the data only for research purposes and not to identify any individual participant;
  * A commitment to protect data through the use of appropiate information technology;
  * A commitment to destroy or return the data after analyses are complete.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data and definitive documentation of the project will be stored centrally on virtual servers (up to 40 TB) and research storage infrastructures provided by the Hospital del Mar Medical Research Institute, during the lifetime of the projects. Thereafter, the data will be kept for the recommended period of 20 years, as set out in the Medical Research Council's guideline "Personal Information in Medical Research" (section 7).
Access Criteria: Data sharing agreement among institutions.

REFERENCES:
- [Background] Zamora V, Garin O, Fumadó Ll, Bonet X, Castells M, Pont A, Gutiérrez C, Ventura M, Ferrer M. Impact of the new treatment modalities in patients with localized prostate cancer. Gac Sanit 2019; 33 Suppl C:224.
- [Background] Sayol L, Garin O, Pont A, Guedea F, Gutiérrez C, Ventura M, Martí-Pastor M, Ferrer M. Men undergoing active surveillance for localized prostate cancer present the best short-term quality of life outcomes. Quality of Life Research 2017;26:1-142 (206.1).
- [Background] Sayol L, Garin O, Pont A, Guedea F, Gutiérrez C, Ventura M, Ferrer M. [Patients under active surveillance with localized prostate cancer are those with the best quality of life in the short-term]. Gaceta Sanitaria 2017;31 (Espec Congr):787.
- [Result] Zamora V, Garin O, Pardo Y, Pont A, Gutierrez C, Cabrera P, Gomez-Veiga F, Pijoan JI, Litwin MS, Ferrer M; Multicentric Spanish Group of Clinically Localized Prostate Cancer. Mapping the Patient-Oriented Prostate Utility Scale From the Expanded Prostate Cancer Index Composite and the Short-Form Health Surveys. Value Health. 2021 Nov;24(11):1676-1685. doi: 10.1016/j.jval.2021.03.021. Epub 2021 Sep 8. PMID 34711369
- [Result] Zamora V, Garin O, Suarez JF, Gutierrez C, Guedea F, Cabrera P, Castells M, Herruzo I, Fumado L, Samper P, Ferrer C, Regis L, Pont A, Ferrer M; Multicentric Spanish Group of Clinically Localized Prostate Cancer. Comparative effectiveness of new treatment modalities for localized prostate cancer through patient-reported outcome measures. Clin Transl Radiat Oncol. 2023 Oct 29;44:100694. doi: 10.1016/j.ctro.2023.100694. eCollection 2024 Jan. PMID 38021091